CLINICAL TRIAL: NCT07019337
Title: Oral Metronomic Capecitabine Combined With Pyrotinib in ADC-treated HER2-positive Metastatic Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ma Fei，MD, Department of Medical Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-112
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: HER2-positive Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pyrotinib plus capecitabine (Experimental): Patients who experienced disease progression (PD) following front-line treatment with an ADC-based regimen received pyrotinib in combination with metronomic capecitabine until disease progression or unacceptable toxicity.
  Interventions: Drug: Pyrotinib; Drug: Capecitabine
- pyrotinib and capecitabine (Experimental): Patients without disease progression who discontinued front-line ADC therapy due to intolerable toxicity, economic reasons, or patient preference were enrolled and received pyrotinib plus metronomic capecitabine until disease progression or unacceptable toxicity.
  Interventions: Drug: Pyrotinib; Drug: Capecitabine

INTERVENTIONS:
Drug: Pyrotinib — 400mg or 320mg qd
Drug: Capecitabine — 500mg tid

SUMMARY:
This is a prospective, open-label, multi-cohort, phase II study to evaluate the efficacy and safety of Oral metronomic capecitabine combined with pyrotinib in patients with HER2-positive advanced breast cancer who had received prior anti-HER2 ADC drugs (including T-DXd, SHR-A1811, T-DM1, etc.) before treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 and ≤75 years.
2. Histologically or cytologically confirmed HER2-positive metastatic breast cancer.
3. Patients must have either experienced disease progression following anti-HER2 antibody-drug conjugate (ADC) therapy in the advanced/metastatic setting (including regimens containing SHR-A1811, T-DXd, T-DM1, or other approved ADCs) or discontinued prior anti-HER2 ADC treatment due to intolerable toxicity, financial constraints, or patient preference without evidence of disease progression.
4. ECOG performance status of 0 to 2.
5. The functions of the main organs are basically normal
6. Signed informed consent

Exclusion Criteria:

1. Prior treatment with a TKI or capecitabine (or other fluoropyrimidine-based chemotherapy) in the advanced or metastatic setting.
2. Known dihydropyrimidine dehydrogenase (DPD) deficiency.
3. Pregnant or lactating patients;
4. Malignancy (except basal cell carcinoma of the skin, which has been cured, and carcinoma in situ of the cervix) in the past 5 years;
5. History of allergic reactions attributed to compounds of similar chemical or biologic composition to the study agent or accompanying supportive medications;
6. Serious physical or mental illnesses or laboratory abnormalities that may increase the risk of participating in the study or interfere with the study results
7. Deemed by the investigator to be ineligible for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | The observation period related to this endpoint is up to 36 months.

SECONDARY OUTCOMES:
Objective response rate (ORR) | The observation period related to this endpoint is up to 36 months.
Clinical Benefit Rate (CBR) | The observation period related to this endpoint is up to 36 months.
Overall Survival (OS) | The observation period related to this endpoint is up to 36 months.
Safety(adverse Events [AEs] and Serious Adverse Events [SAEs]) | From consent through 28 days following treatment completion